CLINICAL TRIAL: NCT01846611
Title: A Randomized, Open-Label Study Comparing the Combination of YONDELIS and DOXIL/CAELYX With DOXIL/CAELYX Monotherapy for the Treatment of Advanced-Relapsed Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: A Study Comparing the Combination of Trabectedin (YONDELIS) and DOXIL/CAELYX With DOXIL/CAELYX for the Treatment of Advanced-Relapsed Epithelial Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100983; ET743OVC3006 (Other: Janssen Research & Development, LLC); 2012-004808-34 (EudraCT Number)
Record Dates: First submitted 2013-05-01; First posted 2013-05-03 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms
Keywords: Ovarian neoplasms; Peritoneal neoplasms; Fallopian tube neoplasms; Advanced-relapsed epithelial ovarian cancer; Advanced-relapsed primary peritoneal cancer; Advanced-relapsed fallopian tube cancer; Trabectedin; Yondelis; Doxil; Caelyx; Platinum sensitive; Tthird-line; BRCA; Patient related outcome
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms | interventions — Trabectedin; liposomal doxorubicin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: trabectedin + DOXIL (Experimental): Participants will receive DOXIL 30 millgram per meter square (mg/m^2) administered as an intravenous (IV) infusion over approximately 90 minutes followed by trabectedin 1.1 mg/m^2 administered as an IV infusion over approximately 3hours, every 3 weeks. Participants will be pretreated with 20 mg dexamethasone IV (or the IV equivalent) approximately 30 minutes before DOXIL study drug. As of Amendment 6, treatment with trabectedin will be discontinued for participants on treatment with trabectedin and no new participants will receive trabectedin. Participants who, in the opinion of the investigator, are deriving clinical benefit may continue treatment with single-agent DOXIL as per the local standard of care.
  Interventions: Drug: Trabectedin; Drug: DOXIL; Drug: Dexamethasone
- Arm B: DOXIL (Active Comparator): Participants will receive DOXIL, 50 mg/m^2 administered as an IV infusion over approximately 90 minutes every 4 weeks.
  Interventions: Drug: DOXIL

INTERVENTIONS:
Drug: Trabectedin — 1.1 mg/m^2 administered intravenously over approximately 3 hours on Day 1 of each 21-day treatment cycle.
  Arms: Arm A: trabectedin + DOXIL
Drug: DOXIL — 30 mg/m^2 administered intravenously over approximately 90 minutes on Day 1 of each 21-day treatment cycle.
  Arms: Arm A: trabectedin + DOXIL
Drug: Dexamethasone — 20 mg administered intravenously on Day 1 of each 21-day treatment cycle approximately 30 minutes prior to study drug infusion.
  Arms: Arm A: trabectedin + DOXIL
Drug: DOXIL — 50 mg/m^2 administered intravenously over approximately 90 minutes on Day 1 of each 28-day treatment cycle.
  Arms: Arm B: DOXIL

SUMMARY:
The purpose of this study is to assess the efficacy and safety of trabectedin+DOXIL as a third-line chemotherapy regimen (treatment) in patients with platinum-sensitive advanced-relapsed epithelial ovarian, primary peritoneal, or fallopian tube cancer who received 2 previous lines of platinum-based chemotherapy.

DETAILED DESCRIPTION:
This is a randomized (individuals assigned to study treatment by chance), open - label (identity of assigned study drug will be known), active - controlled study in adult female patients with platinum-sensitive advanced - relapsed epithelial ovarian, primary peritoneal, or fallopian tube cancer who received 2 previous lines of platinum - based chemotherapy. Approximately 670 participants will be enrolled. Patients will be stratified by 4 criteria defined in the protocol and randomly assigned in a 1:1 ratio to the trabectedin+DOXIL combination therapy group (Arm A) or to the DOXIL (pegylated liposomal doxorubicin) monotherapy group (Arm B). During the treatment phase, patients will receive study drug infusions according to 21 - day cycles in Arm A and 28 - day cycles in Arm B. Treatment will continue until the occurrence of disease progression or unacceptable treatment toxicity, or until 2 cycles after assessment of a complete response (CR). Efficacy assessments will be evaluated using Response Evaluation Criteria in Solid Tumors. Disease assessments, including assessments for patients who discontinue treatment for reasons other than disease progression, will be performed until disease progression, the start of subsequent anticancer therapy, withdrawal of consent, or the clinical cutoff date. Collection of survival status will continue until at least 514 deaths have been observed or until the clinical data cutoff date. Serial pharmacokinetic (PK) samples will be collected in a subset of patients who voluntarily consent to the PK portion of the study. Safety will be monitored throughout the study. An interim analysis of overall survival (OS) will be performed after approximately 308 participants have died. The final analysis of OS will occur when approximately 514 deaths have been observed or until the clinical cutoff date. As of Amendment 6, no new participants will be randomized to study treatment, and treatment with trabectedin should be immediately discontinued for participants assigned to Arm A (trabectedin+DOXIL). All study participants (Arm A or Arm B) currently on study who, in the opinion of the investigator, are deriving clinical benefit may continue treatment with single-agent DOXIL as per the local standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced-relapsed epithelial ovarian, primary peritoneal, or fallopian tube cancer
* Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1
* Received first-line treatment with a platinum-based regimen and had no evidence of disease progression for >= 6 months after the last dose
* Received second-line treatment with a platinum-based regimen, with progression of disease after attaining a response
* Progression of disease based on imaging after the second-line platinum-based regimen (individuals treated with a pegylated liposomal doxorubicin-containing regimen as a second-line therapy are eligible if subsequent disease progression occurs >=9 months from the first dose)
* Evidence of measurable disease at screening as evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) (Version 1.1)
* Participants no longer need to be able to receive intravenous (IV) dexamethasone or an equivalent IV corticosteroid
* Have a known BRCA 1/2 mutation status (for participants who do not have a known BRCA 1/2 status at screening, a blood sample will be collected to determine the status with the results available prior to randomization
* Laboratory values within protocol -defined parameters
* Have left ventricular ejection fraction by multigated acquisition scan (MUGA) scan or 2D-ECHO within normal limits for the institution
* Have side effects (except alopecia) of prior treatment resolved to at least Grade 1 according to the National Cancer Institute - Common Terminology Criteria of Adverse Events (NCICTCAE) (Version 4.0)
* Have a negative urine or serum pregnancy test at screening
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Diagnosis of ovarian carcinoma with mucinous histology
* Had more than 2 prior lines of systemic therapy. Maintenance therapies and hormonal therapies are not considered additional lines of therapy
* Participants who had a prior exposure to trabectedin or hypersensitivity to any of the excipients will not be excluded from receiving single-agent Doxil
* Prior treatment with doxorubicin or other anthracycline at cumulative doses greater than 300 mg/m2 (calculated using doxorubicin equivalent doses: 1 mg doxorubicin = 1 mg Doxil/Caelyx = 1.8 mg epirubicin = 0.3 mg mitoxantrone = 0.25 mg idarubicin)
* Participants unwilling or unable to have a central venous catheter placed will not be excluded from receiving single-agent Doxil
* Pregnant or breast-feeding
* Would receive study treatment within 3 weeks from radiation therapy, experimental therapy, hormonal therapy, prior chemotherapy, or biological therapy; use an invasive investigational device; or is currently enrolled in an investigational study
* History of another invasive malignancy (except non-metastatic basal cell carcinoma or squamous cell carcinoma of the skin or cervical carcinoma in situ adequately treated) unless in remission for >=5 years, or a non - invasive malignancy requiring ongoing therapy
* Known allergies, hypersensitivity, or intolerance to Doxil, dexamethasone, or their excipients
* Known history of central nervous system metastasis
* Known significant chronic liver disease, such as cirrhosis or active hepatitis (potential participants who test positive for hepatitis B surface antigen or hepatitis C antibodies are allowed provided they do not have active disease requiring antiviral therapy)
* Had a myocardial infarct within 6 months before enrollment, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Has any of the following medical conditions: uncontrolled diabetes, psychiatric disorder (including dementia) that prevents compliance with protocol, uncontrolled seizures, newly diagnosed deep vein thrombosis, active systemic infection that is likely to interfere with study procedure or results
* Has any condition that, in the opinion of the investigator, would compromise the well-being of the participant or the study or prevent the participant from meeting or performing study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (138):
- United States (75):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Scottsdale, Arizona
  - Sedona, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Greenbrae, California
  - La Jolla, California
  - Los Angeles, California
  - Orange, California
  - Sacramento, California
  - Englewood, Colorado
  - New Britain, Connecticut
  - New Haven, Connecticut
  - Stamford, Connecticut
  - Fort Myers, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Park Ridge, Illinois
  - Indianapolis, Indiana
  - Louisville, Kentucky
  - Covington, Louisiana
  - New Orleans, Louisiana
  - Scarborough, Maine
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Lansing, Michigan
  - Duluth, Minnesota
  - Edina, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Hackensack, New Jersey
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Summit, New Jersey
  - Brightwaters, New York
  - Hawthorne, New York
  - New York, New York
  - Pinehurst, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Abington, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Austin, Texas
  - Bedford, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas
  - The Woodlands, Texas
  - Webster, Texas
  - Salt Lake City, Utah
  - Annandale, Virginia
  - Newport News, Virginia
  - Roanoke, Virginia
  - Spokane, Washington
  - Vancouver, Washington
  - Green Bay, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
  - Wauwatosa, Wisconsin
- Australia (10):
  - Adelaide
  - Ballarat
  - Brisbane
  - Gosford
  - Parkville
  - Subiaco
  - Toorak Gardens
  - Townsville
  - Wodonga
  - Woodville
- China (4):
  - Guangzhou
  - Jinan
  - Shanghai
  - Shenyang
- Israel (10):
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
  - Ẕerifin
- New Zealand (2):
  - Auckland
  - Wellington
- Poland (5):
  - Bydgoszcz
  - Gdansk
  - Lublin
  - Poznan
  - Warsaw
- Russia (16):
  - Arkhangelsk
  - Chelyabinsk
  - Ivanovo
  - Kirov
  - Krasnodar
  - Moscow
  - Nal'chik
  - Nizhny Novgorod
  - Omsk
  - Orenburg
  - Pyatigorsk
  - Ryazan
  - Saint Petersburg
  - Sochi
  - Ufa
  - Yaroslavl
- South Africa (6):
  - Cape Town
  - Durban
  - eManzimtoti
  - Johannesburg
  - Port Elizabeth
  - Pretoria
- Switzerland (2):
  - Bern
  - Zurich
- United Kingdom (8):
  - Bebington
  - Glasgow
  - Guildford
  - London
  - Maidstone
  - Manchester
  - Plymouth
  - Swansea

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Jones RL, Herzog TJ, Patel SR, von Mehren M, Schuetze SM, Van Tine BA, Coleman RL, Knoblauch R, Triantos S, Hu P, Shalaby W, McGowan T, Monk BJ, Demetri GD. Cardiac safety of trabectedin monotherapy or in combination with pegylated liposomal doxorubicin in patients with sarcomas and ovarian cancer. Cancer Med. 2021 Jun;10(11):3565-3574. doi: 10.1002/cam4.3903. Epub 2021 May 7. PMID 33960681
- [Derived] Monk BJ, Herzog TJ, Wang G, Triantos S, Maul S, Knoblauch R, McGowan T, Shalaby WSW, Coleman RL. A phase 3 randomized, open-label, multicenter trial for safety and efficacy of combined trabectedin and pegylated liposomal doxorubicin therapy for recurrent ovarian cancer. Gynecol Oncol. 2020 Mar;156(3):535-544. doi: 10.1016/j.ygyno.2019.12.043. Epub 2020 Jan 8. PMID 31924332

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 581 participants were enrolled. Out of which 5 participants who were enrolled at the time of study termination were not assigned to any treatment group. Therefore, these 5 participants were not considered as randomized participants and excluded from result analysis.
Groups:
- Trabectedin + DOXIL: Participants received DOXIL 30 milligram per meter square (mg/m^2) administered as an intravenous (IV) infusion over approximately 90 minutes followed by trabectedin 1.1 mg/m^2 administered as an IV infusion over approximately 3 hours, on Day 1 of each treatment cycle (21 days cycle) every 3 weeks. Participants were pretreated with 20 mg dexamethasone IV (or an equivalent IV corticosteroid) approximately 30 minutes prior to initiation of infusion of DOXIL IV.
- DOXIL: Participants received DOXIL 50 mg/m^2 administered as an IV infusion over approximately 90 minutes on Day 1 of each treatment cycle (28 days cycle), every 4 weeks.
Period: Overall Study
Arm/Group | Trabectedin + DOXIL | DOXIL
Started | 289 | 287
Treated | 286 | 282
Completed | 251 | 244
Not Completed | 38 | 43
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 15 | 19
Not completed — Other | 19 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabectedin + DOXIL | DOXIL | Total
Number analyzed (Participants) | 289 | 287 | 576
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (10.16) | 59.9 (10.35) | 59.9 (10.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289 | 287 | 576
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 15
  Not Hispanic or Latino | 270 | 278 | 548
  Unknown or Not Reported | 9 | 4 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 15 | 23 | 38
  Black or African American | 3 | 4 | 7
  Hispanic or Latino | 8 | 3 | 11
  Other | 15 | 11 | 26
  White Non-Hispanic | 248 | 246 | 494
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 15 | 14 | 29
  CHINA | 9 | 18 | 27
  ISRAEL | 2 | 8 | 10
  NEW ZEALAND | 10 | 8 | 18
  POLAND | 3 | 5 | 8
  RUSSIAN FEDERATION | 124 | 122 | 246
  SOUTH AFRICA | 7 | 4 | 11
  SWITZERLAND | 1 | 0 | 1
  UNITED KINGDOM | 15 | 7 | 22
  UNITED STATES | 103 | 101 | 204

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death. Participants who died, regardless of the cause of death, were considered to have had an event.
Time Frame: Up to 4.3 years
Population: All randomized analysis set included all participants who were randomized to study treatment independent of whether they received study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin + DOXIL | DOXIL
Number analyzed (Participants) | 289 | 287
months | 23.82 [20.30 to 26.12] | 22.21 [18.10 to 24.67]
Statistical Analysis 1: Comparison: Trabectedin + DOXIL vs DOXIL; Test type: Superiority; p = 0.5236, Unstratified log rank test; Hazard Ratio (HR) = 0.925, 95% CI 2-sided [0.727 to 1.177]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time between the date of randomization and the date of disease progression or death. PFS was assessed using the response evaluation criteria in solid tumors (RECIST) Version 1.1. As per criteria progressive disease in case of target lesions means at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). Progressive disease in case of non-target lesions means unequivocal progression of existing non-target lesions. In both cases the appearance of one or more new lesions is also considered progression.
Time Frame: Up to 4.3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trabectedin + DOXIL | DOXIL
Number analyzed (Participants) | 289 | 287
months | 7.52 [6.93 to 9.43] | 7.26 [6.14 to 7.59]
Statistical Analysis 1: Comparison: Trabectedin + DOXIL vs DOXIL; Test type: Superiority; p = 0.5174, Unstratified log rank test; Hazard Ratio (HR) = 0.935, 95% CI 2-sided [0.762 to 1.147]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with measurable disease achieving a best overall response of either complete response (CR) or partial response (PR) based on RECIST. CR: disappearance of all target and non-target lesions and normalization of tumor marker levels in non-target lesions. PR: at least a 30 percent (%) decrease in the sum of longest diameter (LD) of target lesions or persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits.
Time Frame: Up to 4.3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Trabectedin + DOXIL | DOXIL
Number analyzed (Participants) | 289 | 287
Percentage of participants | 46.0 [40.2 to 52.0] | 35.9 [30.3 to 41.7]
Statistical Analysis 1: Comparison: Trabectedin + DOXIL vs DOXIL; Test type: Superiority; p = 0.0142, Fisher Exact; Odds Ratio (OR) = 1.523, 95% CI 2-sided [1.075 to 2.158]

ADVERSE EVENTS:
Time Frame: Up to 4.3 years
Description: Safety population included all-treated participants who received at least 1 dose of study drug.
Arm/Group | Trabectedin + DOXIL | DOXIL
All-Cause Mortality (participants affected / at risk) | 132/286 | 131/282
Serious Adverse Events (participants affected / at risk) | 118/286 | 58/282
Other Adverse Events (participants affected / at risk) | 282/286 | 273/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin + DOXIL (N=286) | DOXIL (N=282)
Anaemia (Blood and lymphatic system disorders) | 9 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 14 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 12 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 10 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardiopulmonary Failure (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Inappropriate Antidiuretic Hormone Secretion (Endocrine disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 3
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 3 | 8
Constipation (Gastrointestinal disorders) | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Intestinal Obstruction (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 8 | 3
Neutropenic Colitis (Gastrointestinal disorders) | 0 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 1
Oral Pruritus (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 4 | 14
Stomatitis (Gastrointestinal disorders) | 0 | 2
Subileus (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 10 | 7
Asthenia (General disorders) | 0 | 1
Catheter Site Inflammation (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 0 | 1
Chest Pain (General disorders) | 0 | 1
Death (General disorders) | 4 | 2
Fatigue (General disorders) | 4 | 1
Influenza Like Illness (General disorders) | 1 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 2 | 1
Oedema Peripheral (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 9 | 3
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 2 | 0
Abdominal Wall Abscess (Infections and infestations) | 0 | 1
Catheter Site Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Device Related Infection (Infections and infestations) | 3 | 1
Device Related Sepsis (Infections and infestations) | 1 | 0
Enterobacter Bacteraemia (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 2 | 1
Oral Candidiasis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 2 | 0
Peritonitis Bacterial (Infections and infestations) | 1 | 0
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 4 | 0
Pseudomonal Sepsis (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 4 | 2
Septic Shock (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 5 | 1
Anastomotic Ulcer (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal Stoma Complication (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 2
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 14 | 0
Aspartate Aminotransferase Increased (Investigations) | 9 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 0
Ejection Fraction Decreased (Investigations) | 2 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 5 | 0
Platelet Count Decreased (Investigations) | 3 | 0
Transaminases Increased (Investigations) | 1 | 0
Weight Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Lymphangiosis Carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Abdominal Wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 0
Device Malfunction (Product Issues) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 4 | 2
Renal Failure (Renal and urinary disorders) | 1 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Pelvic Fluid Collection (Reproductive system and breast disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Capillary Leak Syndrome (Vascular disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 3 | 0
Embolism (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Pelvic Venous Thrombosis (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trabectedin + DOXIL (N=286) | DOXIL (N=282)
Anaemia (Blood and lymphatic system disorders) | 135 | 70
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 | 2
Leukopenia (Blood and lymphatic system disorders) | 53 | 38
Neutropenia (Blood and lymphatic system disorders) | 149 | 104
Thrombocytopenia (Blood and lymphatic system disorders) | 63 | 18
Palpitations (Cardiac disorders) | 7 | 6
Tachycardia (Cardiac disorders) | 9 | 2
Vertigo (Ear and labyrinth disorders) | 6 | 6
Abdominal Distension (Gastrointestinal disorders) | 20 | 15
Abdominal Pain (Gastrointestinal disorders) | 54 | 44
Abdominal Pain Lower (Gastrointestinal disorders) | 6 | 7
Abdominal Pain Upper (Gastrointestinal disorders) | 12 | 8
Ascites (Gastrointestinal disorders) | 12 | 17
Constipation (Gastrointestinal disorders) | 82 | 61
Diarrhoea (Gastrointestinal disorders) | 59 | 47
Dry Mouth (Gastrointestinal disorders) | 5 | 10
Dyspepsia (Gastrointestinal disorders) | 23 | 18
Dysphagia (Gastrointestinal disorders) | 1 | 8
Flatulence (Gastrointestinal disorders) | 7 | 8
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 12 | 15
Mouth Ulceration (Gastrointestinal disorders) | 6 | 14
Nausea (Gastrointestinal disorders) | 212 | 114
Oral Pain (Gastrointestinal disorders) | 5 | 10
Stomatitis (Gastrointestinal disorders) | 52 | 91
Vomiting (Gastrointestinal disorders) | 141 | 54
Asthenia (General disorders) | 39 | 16
Chills (General disorders) | 8 | 5
Fatigue (General disorders) | 171 | 113
Malaise (General disorders) | 7 | 5
Mucosal Inflammation (General disorders) | 22 | 33
Non-Cardiac Chest Pain (General disorders) | 11 | 8
Oedema Peripheral (General disorders) | 32 | 22
Pain (General disorders) | 11 | 5
Peripheral Swelling (General disorders) | 9 | 6
Pyrexia (General disorders) | 38 | 26
Pneumonia (Infections and infestations) | 5 | 8
Sinusitis (Infections and infestations) | 5 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 14 | 6
Urinary Tract Infection (Infections and infestations) | 12 | 15
Viral Upper Respiratory Tract Infection (Infections and infestations) | 7 | 11
Contusion (Injury, poisoning and procedural complications) | 8 | 3
Alanine Aminotransferase Increased (Investigations) | 151 | 12
Aspartate Aminotransferase Increased (Investigations) | 100 | 11
Bilirubin Conjugated Increased (Investigations) | 24 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 73 | 16
Blood Bilirubin Increased (Investigations) | 24 | 3
Blood Creatine Phosphokinase Increased (Investigations) | 13 | 9
Blood Creatinine Increased (Investigations) | 20 | 21
Blood Urea Increased (Investigations) | 6 | 4
Ejection Fraction Decreased (Investigations) | 20 | 10
Gamma-Glutamyltransferase Increased (Investigations) | 13 | 5
Haemoglobin Decreased (Investigations) | 6 | 1
Lymphocyte Count Decreased (Investigations) | 8 | 4
Neutrophil Count Decreased (Investigations) | 52 | 37
Platelet Count Decreased (Investigations) | 52 | 16
Weight Decreased (Investigations) | 13 | 16
White Blood Cell Count Decreased (Investigations) | 33 | 29
Decreased Appetite (Metabolism and nutrition disorders) | 83 | 52
Dehydration (Metabolism and nutrition disorders) | 21 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 19 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 24 | 15
Bone Pain (Musculoskeletal and connective tissue disorders) | 11 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 8 | 2
Joint Swelling (Musculoskeletal and connective tissue disorders) | 6 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 16 | 9
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 8 | 16
Dizziness (Nervous system disorders) | 7 | 6
Dizziness Postural (Nervous system disorders) | 10 | 3
Dysgeusia (Nervous system disorders) | 35 | 20
Headache (Nervous system disorders) | 38 | 29
Neuropathy Peripheral (Nervous system disorders) | 11 | 13
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 7
Anxiety (Psychiatric disorders) | 18 | 8
Depression (Psychiatric disorders) | 8 | 14
Insomnia (Psychiatric disorders) | 19 | 16
Pollakiuria (Renal and urinary disorders) | 3 | 7
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 34
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 28
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 10 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16 | 17
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 32 | 22
Dry Skin (Skin and subcutaneous tissue disorders) | 22 | 21
Erythema (Skin and subcutaneous tissue disorders) | 3 | 7
Night Sweats (Skin and subcutaneous tissue disorders) | 5 | 6
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 58 | 117
Pigmentation Disorder (Skin and subcutaneous tissue disorders) | 5 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 14
Rash (Skin and subcutaneous tissue disorders) | 22 | 26
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 8 | 24
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 10 | 12
Skin Toxicity (Skin and subcutaneous tissue disorders) | 3 | 6
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 6
Hot Flush (Vascular disorders) | 7 | 8
Hypertension (Vascular disorders) | 22 | 7
Hypotension (Vascular disorders) | 11 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT01846611/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT01846611/SAP_001.pdf